CLINICAL TRIAL: NCT04513743
Title: Sleep in the Ultra Long-Term Perspective: Seasonality and Behaviorally Induced Variation
Brief Title: Ultra Long-Term Sleep Monitoring Using UNEEG™ Medical 24/7 EEG™ SubQ
Acronym: ULTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNEEG Medical A/S (Industry)
Collaborators: Zealand University Hospital (Other); Cambridge Cognition Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: U003
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Sleep
Keywords: Circadian; Chronobiology; Sleep quality; Automated sleep staging; Implantable device
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy adults (Experimental): UNEEG™ medical 24/7 EEG™ SubQ
  Interventions: Diagnostic Test: 24/7 EEG™ SubQ

INTERVENTIONS:
Diagnostic Test: 24/7 EEG™ SubQ — 24/7 EEG™ SubQ device will be worn by each subject for 365 nights

SUMMARY:
This study aims to evaluate the agreement between automated sleep analysis by UNEEG medical's 24/7 EEG™ SubQ device using a deep learning algorithm and the consensus score of multiple sleep technologists' manual scoring of 120 gold-standard polysomnograms (PSG) from healthy subjects.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the agreement between automated sleep analysis by UNEEG medical's 24/7 EEG™ SubQ device using a deep learning algorithm and the consensus score of multiple sleep technologists' manual scoring of 120 gold-standard polysomnograms (PSG).

The study will enroll 20 healthy subjects who will wear the UNEEG™ SubQ device for 365 consecutive nights. All subjects are prescreened and invited to an interview to confirm eligibility. Subjects who provide informed consent are enrolled and will complete a detailed demographic, medical, health, sleep, and lifestyle survey. The enrolled subjects will have the UNEEG™ SubQ implanted and after approximately 10 days of healing the study subjects will start wearing the external part of the 24/7 EEG™ SubQ. Throughout the study the subjects will wear an ActiGraph, fill out a sleep diary and conduct cognitive tests. The duration of the study from screening to removal of sutures will be approximately 58 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Subjects must be of general good health

Exclusion Criteria:

* Has cochlear implants.
* Involved in therapies with medical devices that deliver electrical energy into the area around the implant
* Is at high risk of surgical complications, such as active systemic infection and hemorrhagic disease.
* Are unable (i.e. mentally or physically impaired patient), or do not have the necessary assistance, to properly operate the device system.
* Has an infection at the site of device implantation.
* Operates MRI scanners.
* Has a profession/hobby that includes activity imposing extreme pressure variations (e.g. diving or parachute jumping). N.B.: diving/snorkeling is allowed to 5 meters depth.
* Has a profession/hobby that includes activity imposing an unacceptable risk for trauma against the device or the site of implantation (e.g. martial art or boxing).
* Previous stroke or cerebral hemorrhage and any other structural cerebral disease.
* Ongoing or history of sleep disorders.
* Known neurological diseases.
* Known or suspected abuse of alcohol defined as estimated consumption beyond that, which is recommended by the Danish Health Authority or any other neuro-active substances.
* Other known diseases or conditions, judged by investigator to influence sleep to such a degree that data quality will be compromised.
* Medication judged by investigator to influence sleep to such a degree that data quality will be compromised.
* Incapable, judged by the investigator, of understanding the participant instruction or who are not capable of carrying through the investigation.
* Pregnancy or intention to become pregnant within the next 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-07-04 (Actual)

PRIMARY OUTCOMES:
Sleep stage agreement | 1 year
  Automatically determined sleep stages using data from 24/7 EEG SubQ, sleep stages manually determined according to the American Academy of Sleep Medicine (AASM) manual using the PSG recordings. The goal is to evaluate the performance of classification of AASM sleep stages at each 30-sec epoch determined automatically from the data recorded using the 24/7 EEG SubQ, to those determined by the consensus score (most prevalent score) of the sleep technologists' scoring of each subject's PSG record from the same night.

SECONDARY OUTCOMES:
Quantitative sleep parameters agreement | 1 year
  The quantitative sleep parameters recommended by the AASM manual. The goal is to evaluate the agreement between automatically determined clinically relevant parameters using data recorded from the 24/7 EEG SubQ and to those determined by the consensus score (most prevalent score) of the sleep technologists' scoring of each subject's PSG record from the same night.
Non-Inferiority in sleep/wake monitoring | 1 year
  Automatically determined sleep/wake epochs using data from 24/7 EEG SubQ, automatically determined sleep/wake epochs using ActiLife 6 and data from ActiGraph Link GT9X, sleep/wake epochs manually determined according to the AASM manual using the PSG recordings. The goal is to show non-inferiority of sleep/wake monitoring using 24/7 EEG SubQ in a head-to-head comparison with actigraphy using PSG as a reference and gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Troels W Kjær, Professor, Principal Investigator — Zealand University Hospital
Locations (1):
- Zealand University Hospital, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahrens E, Jennum P, Duun-Henriksen J, Djurhuus B, Homoe P, Kjaer TW, Hemmsen MC. Automatic sleep staging based on 24/7 EEG SubQ (UNEEG medical) data displays strong agreement with polysomnography in healthy adults. Sleep Health. 2024 Dec;10(6):612-620. doi: 10.1016/j.sleh.2024.08.007. Epub 2024 Oct 15. PMID 39406630